CLINICAL TRIAL: NCT05573529
Title: Comparison of Visual Outcomes and Patient Satisfaction After Bilateral Implantation of EDOF and Multifcoal IOLs- a Prospective Randomized Controlled Trial
Brief Title: EDOF and Multifocal IOL Study
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Medical University of Vienna (Other)
Responsible Party: Principal Investigator, Christina Leydolt, Assoc. Prof. PD Dr, Medical University of Vienna
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 1163/2020
Record Dates: First submitted 2022-09-09; First posted 2022-10-10 (Actual); Last update posted 2025-06-18 (Actual); Status verified 2025-06

CONDITIONS: Age-related Cataract
MeSH Terms: interventions — Phacoemulsification; Lens Implantation, Intraocular

STUDY DESIGN:
Intervention Model Description: intra-individual comparison of two groups recieving predefined EDOF and multifocal intraocular lenses. In group one (I), the EDOF lens one (I) will be implanted in the dominant eye and the multifocal lens one (I) in the non-dominant eye. Subsequently, study participants in group two (II) will receive the EDOF lens one (I) in the dominant eye and the multifocal lens two (II) in the non-dominant eye.
Who Masked: Outcomes Assessor
Masking Description: outcome assessor will be masked to the intraocular lens implanted.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Edof IOL vs. multifocal IOL I (Experimental): The investigational devices are approved intraocular lenses (IOLs) intended to be implanted after phacoemulsification in individuals suffering from age-related cataract with the need of cataract surgery. In Arm one (I) participants will receive Edof IOL one (I) vs. multifocal IOL one (I).
  Interventions: Procedure: phacoemulsification and intraocular lens implantation; Device: intraocular lens implantation
- Edof IOL vs. multifocal IOL II (Experimental): The investigational devices are approved intraocular lenses (IOLs) intended to be implanted after phacoemulsification in individuals suffering from age-related cataract with the need of cataract surgery. In Arm two (II) participants will receive Edof IOL one (I) vs. multifocal IOL two (II).
  Interventions: Procedure: phacoemulsification and intraocular lens implantation; Device: intraocular lens implantation

INTERVENTIONS:
Procedure: phacoemulsification and intraocular lens implantation — bilateral cataract surgery including phacoemulsification in individuals suffering from age-related cataract and intraocular lens implantation
Device: intraocular lens implantation — intraocular lens implantation includes EDOF IOL implantation in the dominant eye and multifocal IOL implantation in the non-dominant eye after phacoemulsification

SUMMARY:
The investigational devices are approved intraocular lenses (IOLs) intended to be implanted after phacoemulsification in individuals suffering from age-related cataract with the need of cataract surgery. Cataract surgery with precedent bilateral randomized IOL implantation will be performed in subjects who have signed an informed consent form. Postoperative examinations will be implemented in accordance with the approved investigational plan.

ELIGIBILITY:
Inclusion Criteria:

* Bilateral age-related cataract for which phacoemulsification extraction and posterior IOL implantation has planned
* Age 50-90
* Visual potential in both eyes of 20/30 or better as determined by investigators estimation
* Normal findings in medical history and physical examination unless the investigator considers an abnormality to be clinically irrelevant

Exclusion Criteria:

* Preceding ocular surgery or trauma
* Relevant other ophthalmic diseases (such as retinal degenerations, etc.)
* Uncontrolled systemic or ocular disease

Ages: 50 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 50 (Actual)
Dates: Start 2020-11-09 (Actual); Primary Completion 2023-03-23 (Actual); Study Completion 2025-02-05 (Actual)

PRIMARY OUTCOMES:
distant corrected near visual acuity | 6 months
  Primary outcome measure will be monocular distant corrected near visual acuity (DCNVA) of each intraocular lens implanted. DCNVA will be assessed using standardized early treatment diabetic retinopathy study (EDTRS) charts on a logarithm of the minimum angle of resolution (logMAR) scale.

OTHER OUTCOMES:
Binocular Uncorrected Near Visual Acuity | 3 years
  Other outcome measure will be binocular uncorrected near visual acuity (UNVA) of each mix-and-match group. Binocular UNVA will be assessed using standardized early treatment diabetic retinopathy study (EDTRS) charts on a logarithm of the minimum angle of resolution (logMAR) scale.

CONTACTS AND LOCATIONS:
Locations (1):
- Medical University of Vienna, Vienna, Vienna, Austria

IPD SHARING:
Plan to Share IPD: Undecided